CLINICAL TRIAL: NCT05982145
Title: The Use of Compression in Institutions and at People's Homes: A Satisfaction Study, Representations, Opinions and Expectations of Users and Caregivers and Creation of a Morphological Database. A Qualitative and Quantitative Multicentric Study
Brief Title: The Use of Compression in Institutions and at People's Homes
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Sigvaris Corporation (Industry); Gerontopole Auvergne Rhone-Alpes (AURA) (Other)
Responsible Party: Sponsor
Other Study IDs: GA-2021-04
Record Dates: First submitted 2021-08-05; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2021-08

CONDITIONS: Aging
Keywords: Compression; Vein
MeSH Terms: interventions — Focus Groups; Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients who are 60 years old and over: Patients who are 60 years old and over had a questionary and a measure of their leg's length
  Interventions: Other: Questionary and measures
- Patients with / or had venous leg ulcers: Patients with / or had venous leg ulcers actually have individual interviews
  Interventions: Other: Individual interviews
- Caregivers who treat patients with venous leg ulcers (except nursing homes): Caregivers who treat patients with venous leg ulcers (except nursing homes) actually have individual interviews
  Interventions: Other: Individual interviews
- Caregivers in nursing homes for dependant elderly people and institutions like hospital: Caregivers in nursing homes for dependant elderly people and institutions like hospital actually have focus groups
  Interventions: Other: Focus groups

INTERVENTIONS:
Other: Individual interviews — Identify the needs and expectations of the users about the compression therapy; Identify the possible facilities and difficulties in link with the management of the venous leg ulcers; Identify care experiences; Identify experiences about the actual compressions systems
  Groups: Caregivers who treat patients with venous leg ulcers (except nursing homes); Patients with / or had venous leg ulcers
Other: Focus groups — Identify facilities and difficulties in link with the prescription and implementation of the compression therapy everyday
  Groups: Caregivers in nursing homes for dependant elderly people and institutions like hospital
Other: Questionary and measures — To take measurement of patients who lives in institution or at their home and take measure of hydration and some other measures like the Group Iso Resource (GIR) and the capacity of the person to getting out of the bed.
  Groups: Patients who are 60 years old and over

SUMMARY:
The compression therapy is a main treatment for chronic venous disease and its different phases. It has proven its effectiveness and usefulness in preventive phase and curative phase. Gérontopôle AURA leads with his partner Sigvaris a large study about the compression in institutions and at patient's homes. Indeed, through 3 studies, the mains goals are to identify the facilities and difficulties about the use of the actual tools. The final aim is to propose a future compression device wich could be adapted and that responds to the needs of users and the realities of the field. First study: Construction of a representative morphological database of people who are 60 years old and older. Indeed, the actually sizing tables are not specifics so not adapted to the morphology of the wearer. This can have an impact on the effectiveness of the treatment and the comfort of the patient. Second study: Have a deep comprehension about the pathway of the compression stockings and bandage in public and private establishment specifically retirements homes for dependant elderly people and hospital. The objectives are to understand and identify the role of health professionals from prescription to implementation to the compressive tools and have their feeds backs. Moreover, the goal is to collect the uses and constraints related to compression systems and to identify the possible improvements, needs and hindrances in link with compressions products. Third study: Study of acceptability of a new adjustable compression solution for venous ulcers. The main goal is to understand the needs and expectations by the users and to know if a new adjustable compression system could be accepted by them. For that, it's important to have a feed back about the use of the compression by the caregivers, medical staff and patients and evaluate the comfort about the use of the compression at patient's home and in institutions. Getting their advices, opinions are necessary too.

DETAILED DESCRIPTION:
The mains goals are to identify the facilities and difficulties about the use of the actual tools. The final aim is to propose a future compression device wich could be adapted and that responds to the needs of users and the realities of the field.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 :

Patients who are 60 years old and over Patients who have or not a compression therapy Patients who have a social security system Patients who have received information of the study and who approbate their participation

- Group 2 et 3 : People who have or had venous leg ulcers People who use or have used compression therapy People who can understand and exchange with the researcher People who have received information of the study and who approbate their participation

- Group 4 : Professionals who work in the investigated institution Professionals who have a link with patients who have a compression therapy Professionals who have received information of the study and who approbate their participation

Exclusion Criteria:

* Group 1 :

Patients who refused to participate at the study Patients who are under 60 years old.

- Group 2 et 3 : People with cognitive disorders People who have no link with venous leg ulcers People who have or had wounds except venous leg ulcers People who refused to participate

- Group 4 : Professionals who have no link with patients who have compression therapy Profession who refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group 1 : People who are 60 years old and older
  * Group 2 : Patients who had or have venous leg ulcers
  * Group 3 : Caregivers who work near and treat patients with venous leg ulcers
  * Group 4 : Caregivers in nursing homes and institutions like hospital
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
data about leg's length | Months 5
  Collect representative data about leg's length. Measure by questionary and taking measures
data about measure of hydration | Months 5
  Collect representative data about measure of hydration. Measure by questionary and taking measures
data about the Group Iso Resource (GIR) | Months 5
  Collect representative data about the Group Iso Resource (GIR). Measure by questionary and taking measures
data about the capacity of the person to getting out of the bed. | Months 5
  Collect representative data about the capacity of the person to getting out of the bed. Measure by questionary and taking measures

SECONDARY OUTCOMES:
caregivers's experiences and representations about compression systems of venous leg ulcer | Months 6
  Measure by individuals interviews
patients' experiences and representations about compression systems of venous leg ulcer | Months 6
  Measure by individuals interviews

OTHER OUTCOMES:
caregivers's in institution experiences and representations about the pathway of compression systems in institution | Months 18
  Measure by Focus Groups

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Barth, PHD, Study Chair — Gerontopole Auvergne Rhone-Alpes (AURA)
Locations (1):
- Gérontopole AURA, Saint-Etienne, France